CLINICAL TRIAL: NCT05652907
Title: A Randomized, Double-Blind Placebo Controlled Parallel Group Study of Safety and Efficacy of FSD201 in Patients With Chronic Widespread Musculoskeletal Nociplastic Pain Associated With Idiopathic Mast Cell Activation Syndrome (Disorder)
Brief Title: Safety and Efficacy of FSD201 for the Treatment of Chronic Pain Associated With Idiopathic MCAS (MCAD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: For business reasons and not for reasons related to safety or efficacy
Sponsor: Quantum Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FSD201-010
Record Dates: First submitted 2022-11-23; First posted 2022-12-15 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-02

CONDITIONS: Mast Cell Activation Syndrome; Mast Cell Activation Disorder Idiopathic
MeSH Terms: conditions — Mast Cell Activation Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FSD201 (Experimental): Participants will receive 600 milligrams (mg) FSD201 tablet twice daily (BID) orally from Day 0 to Day 56.
  Interventions: Drug: FSD201
- Placebo (Placebo Comparator): Participants will receive placebo matched to 600 mg FSD201 tablets twice daily (BID) orally from Day 0 to Day 56.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FSD201 — Tablets for oral administration.
  Arms: FSD201
Drug: Placebo — Placebo tablets matched to FSD201 for oral administration.
  Arms: Placebo

SUMMARY:
This study will determine if FSD201 reduces the average daily 24-hour recall pain intensity after 28 and 56 days of treatment in adults with chronic widespread musculoskeletal nociplastic pain.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of idiopathic MCAS as per the global consensus diagnostic criteria
* Adults with widespread chronic pain (in three or more body regions);
* Chronic pains of intensity greater than or equal to 4.0 but less than or equal to 9.0 on a Numeric Pain Rating Scale, symptom duration of more than 6 months;
* Subject agrees to use only acetaminophen (up to 1000 mg per dose and not to exceed 3000 mg/day) or diphenhydramine (up to 300 mg/day) as rescue medication for chronic widespread musculoskeletal nociplastic pains throughout the trial;
* The subject is willing to maintain current activity and exercise levels throughout the study;
* During the study, the subject agrees not to initiate or change any non-pharmacologic interventions (including chiropractic care, physical therapy, psychotherapy, and massage therapy). Any ongoing non-pharmacologic intervention must be stable for at least 4 weeks before screening and should be continued for the duration of the study;

Key Exclusion Criteria:

* The subject has pain that cannot be clearly differentiated from or that could interfere with the assessment of chronic musculoskeletal nociplastic pain secondary likely to idiopathic MCAS (post-herpetic neuralgia, traumatic injury, prior surgery, complex regional pain syndrome);
* Adults with chronic cancer pain;
* Adults with inflammatory connective tissue disorder or rheumatological disorder-related pain, for example rheumatoid arthritis;
* Adults with focal musculoskeletal pain;
* Adults with skin diseases (chronic urticaria, pemphigus, lupus, rosacea etc.);
* Adults with endocrinological disorders (acute hypothyroidism, acute adrenal insufficiency etc.);
* Adults with systemic gastrointestinal conditions (Inflammatory bowel disorders);
* Significant psychological comorbidities: PHQ-9 score greater than 20; and GAD-7 score greater than 15 (indication of severe anxiety that could interfere with accurate logging of pain ratings);
* Current or recent (within 12 months of screening) history of a substance use disorder including cannabinoid or alcohol use disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders (5th edition; DSM-5);
* Subject has neurologic disorder unrelated to chronic widespread musculoskeletal nociplastic pains (phantom limb from amputation, vitamin B12 deficiency, chronic inflammatory demyelinating polyneuropathy), circulatory disorder (peripheral artery disease), a skin condition in the area of neuropathy that could alter sensation (plantar ulcer), or other painful conditions (arthritis) that could interfere with reporting of pain due to chronic widespread musculoskeletal nociplastic pains;
* Current severe or uncontrolled major depressive disorder or anxiety disorders. Mild to moderate major depression or anxiety disorders are permitted provided that the investigator assesses the patient as clinically stable and appropriate for entry into the study. Stable doses of SSRIs are allowed for the treatment of depression if the dose is stable for 60 days before Screening Visit;
* Subject has a history of suicide attempt or suicidal behaviour within the last 12 months or has suicidal ideation within the previous 12 months or who is at significant risk to commit suicide, as judged by the Investigator at Screening and/or Randomization Visit;
* Patients with active malignancy or history of malignancy, except for basal cell or squamous cell carcinoma and actinic keratosis. Basal cell carcinoma and small squamous cell carcinoma of the skin which have been excised according to guidelines within the last 5 years or in situ cervical carcinoma that has been fully treated and shows no evidence of recurrence are allowed;
* Individuals with generalized joint hypermobility secondary to hereditary connective tissue disorders like Ehlers Danlos Syndrome;
* Individuals with high baseline serum tryptase levels suggestive of Primary or Secondary MCAS (defined as above the normal range of 2.2 to 13.2 µg/L).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Targeted treatment effect of 30% decrease from baseline to Day 28 in the average daily pain intensity | Day 28
  Targeted treatment effect of 30% decrease from baseline to Day 28 in the average daily pain intensity score measured by an 11-point numerical pain rating scale (NPRS). NPRS is an 11-point scale from 0 to10 where the higher number indicates worse pain.
  Averages will be calculated as follows: Baseline: calculated weekly average from Day -7 to Day -1 Day 28: calculated weekly average from Day 22 to Day 28

SECONDARY OUTCOMES:
Percentage of subjects achieving ≥30% reduction in Numerical Pain Rating Scale (NPRS) score at the end of treatment with FSD201 at the end of treatment with FSD201 | Day 28, Day 56
  Change from baseline in the weekly average of the average daily pain intensity measured by Numerical Pain Rating Scale (NPRS). NPRS is an 11-point scale from 0 to 10 where the higher number indicates worse pain.
  NPRS averages will be calculated as follows: Baseline: calculated weekly average from Day -7 to Day -1 Day 28: calculated weekly average from Day 22 to Day 28 Day 56: calculated weekly average from Day 49 to Day 55 for the NPRS.
Change in Patient Global Impression of Change (PGIC) | Day 56
  Change in Patient Global Impression of Change (PGIC) after 56 days treatment from 1 to 7 where the higher number indicates a larger improvement.
Change or reduction in patient average daily NPRS | Day 56
  Change or reduction in patient average daily Numerical Pain Rating Scale (NPRS) after 56 days treatment. NPRS is an 11-point scale from 0 to 10 where the higher number indicates worse pain.
  NPRS averages will be calculated as follows: Baseline: calculated weekly average from Day -7 to Day -1 Day 56: calculated weekly average from Day 49 to Day 55 for the NPRS
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance- Short Form (SF) 8a | Day 56
  Change from baseline (Day 0) in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance - Short Form (SF) 8a after 56 days treatment. PROMIS sleep disturbance is a series of 8 questions, each on a 5-point scale (1-5) where the higher number indicates a worse outcome. A total score out of 40 will be calculated.
Change in the PROMIS Pain Interference- SF 8a score | Day 56
  Change from baseline (Day 0) in the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference - SF 8a score after 56 days treatment. PROMIS pain interference is a series of 8 questions, each on a 5-point scale (1-5) where the higher number indicates a worse outcome. A total score out of 40 will be calculated.
Change in the PROMIS General Life Satisfaction- SF 5a | Day 56
  Change from baseline (Day 0) in the Patient-Reported Outcomes Measurement Information System (PROMIS) General Life Satisfaction - SF 5a after 56 days treatment. PROMIS General Life Satisfaction is series of 5 questions, each on a 7-point scale (1-7) where the higher number indicates a better outcome. A total score out of 35 will be calculated.
Change in the PROMIS Fatigue- SF 8a | Day 56
  Change from Baseline (Day 0) in the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue - SF 8a after 56 days treatment. PROMIS Fatigue is a series of 8 questions, each on a 5-point scale (1-5) where the higher number indicates a worse outcome. A total score out of 40 will be calculated.
Reduction of plasma serum mast cell tryptase, IL-6, and IL-1beta during FSD201 treatment | Day 14, Day 28 and Day 56
  Determine whether FSD201 treatment reduces serum mast cell tryptase, IL6, and IL-1beta during treatment compared to Day 0
Percentage of subjects achieving ≥30% reduction in NPRS score | Day 28, Day 56
  Percentage of subjects achieving ≥30% reduction in Numerical Pain Rating Scale (NPRS) score. NPRS is an 11-point scale from 0 to10 where the higher number indicates worse pain.
  NPRS averages will be calculated as follows: Baseline: calculated weekly average from Day -7 to Day -1 Day 28: calculated weekly average from Day 22 to Day 28 Day 56: calculated weekly average from Day 49 to Day 55 for the NPRS
Change in Daily Sleep Interference Scale (DSIS) | Day 28, Day 56
  Daily Sleep Interference Scale (DSIS) is an 11-point scale (0-10 where the higher number indicates worse ability to sleep.
  Averages will be calculated as follows: Baseline: calculated weekly average from Day -7 to Day -1 Day 28: calculated weekly average from Day 22 to Day 28 Day 56: calculated weekly average from Day 50 to Day 56 for the DSIS
Change in Patient Global Impression of Change (PGIC) | Day 28, Day 56
  Change in Patient Global Impression of Change (PGIC) from 1 to 7 where the higher number indicates a larger improvement.
Change in pain intensity on the NPRS from baseline to each week of treatment | Day 0 to Day 56
  Change in pain intensity on the Numerical Pain Rating Scale (NPRS) score from baseline to each week of treatment. NPRS is an 11-point scale from 0 to 10 where the higher number indicates worse pain.
  Averages will be calculated as follows: Baseline: calculated weekly average from Day -7 to Day -1; Week 1: calculated weekly average from Day 0 to Day 6; Week 2: calculated weekly average from Day 7 to Day 13; Week 3: calculated weekly average from Day 14 to Day 20; Week 4: weekly average from Day 21 to Day 27; Week 5: calculated weekly average from Day 28 to Day 34; Week 6: calculated weekly average from Day 35 to Day 41; Week 7: calculated weekly average from Day 42 to Day 48; Week 8: calculated weekly average from Day 49 to Day 55
Percentage of subjects achieving ≥50% reduction in NPRS | Week 1 to Week 8
  Change from baseline in the weekly average of the average daily pain intensity measured by Numerical Pain Rating Scale (NPRS) score from baseline to each week of treatment. NPRS is an 11-point scale from 0 to 10 where the higher number indicates worse pain.
  Baseline: calculated weekly average from Day -7 to Day -1 Day 56: calculated weekly average from Day 49 to Day 55
Total amount of rescue medication used | Day 0 to Day 56
  Total amount of rescue medication used
Incidence and severity of treatment-emergent adverse events (TEAEs) | Day 0 to Day 56
  Incidence and severity of treatment-emergent adverse events (TEAEs) throughout the dosing period
Incidence and severity of treatment-emergent changes in laboratory values | Day 56
  Incidence and severity of treatment-emergent changes in laboratory values at Day 56
Change from baseline in sitting blood pressure at each in-patient visit | Day 14, Day 28, Day 56
  Change from baseline (Day 0) in sitting blood pressure at each in-patient visit
Change from baseline in heart rate at each in-patient visit | Day 14, Day 28, Day 56
  Change from baseline (Day 0) in heart rate at each in-patient visit
Change from baseline in body temperature at each in-patient visit | Day 14, Day 28, Day 56
  Change from baseline (Day 0) in body temperature at each in-patient visit
Change from baseline in oxygen saturation at each in-patient visit | Day 14, Day 28, Day 56
  Change from baseline (Day 0) in oxygen saturation using Pulse oximetry at each in-patient visit
Change from baseline in breathing rate at each in-patient visit | Day 14, Day 28, Day 56
  Change from baseline (Day 0) in breathing rate at each in-patient visit

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Chruscinski, MD, Study Director — FSD Pharma
Locations (3):
- United States (2):
  - Saint Charles Clinical Research, Weldon Spring, Missouri
  - Norman Marcus Pain Institute, New York, New York
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No